CLINICAL TRIAL: NCT00641810
Title: The Effect of Caffeine Reduction on Snoring and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Benjamin Littenberg, Professor of Medicine, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-123
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Snoring
Keywords: Caffeine; Snoring; Sleep
MeSH Terms: conditions — Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): After one week at usual levels of caffeine use, patients are asked to reduce their caffeine consumption to no more than 2 cups of coffee (or equivalent) for one week and then to zero for two weeks.
  Interventions: Behavioral: Caffeine reduction

INTERVENTIONS:
Behavioral: Caffeine reduction — Reduction in daily caffeine consumption from usual amounts to none.

SUMMARY:
Snoring is a problem for many people, often disturbing energy level, quality of sleep, and the relationship with a bed partner. Two observational studies that have indicated a relationship between the consumption of caffeine and snoring. The objective of this study will be to observe the degree of snoring and quality of sleep when caffeine intake is reduced over a period of four weeks. This will be a prospective, before-and-after study of a behavioral intervention.

This study will engage thirty adults who report snoring, drink two cups of coffee or more per day (or an equivalent amount of caffeine), and have a consistent bed partner who can report on snoring severity. Both subject and partner will be asked to fill out a diary each day. The subjects will record the type of caffeine consumed, time at which each beverage was ingested, the total minutes of physical exercise, any caffeine withdrawal symptoms, quality of sleep, and energy in the morning. The partner (reporter) will rate his or her own sleep quality and energy in the morning, as well as the snoring level of the subject. Beginning the second week of the study, the subject will reduce caffeine intake to half the baseline consumption, and on the third week, will eliminate caffeine altogether.

At the end of each week, the participants will be asked to mail their diaries in to the researchers and start a new series of entries. The study team will also call each week to answer any questions or concerns of the subject and reporter, and encourage continued reporting. When six weeks have elapsed following the completion of the last diary, the investigators will make a final call to the participants to record their current level of snoring, quality of sleep, and daily energy level.

ELIGIBILITY:
Inclusion Criteria:

* age at least 18 years
* consume 16 ounces of coffee or 25 ounces of caffeinated soda or tea
* consistent bed partner willing to serve as reporter
* reported as a loud snorer (6 or more on 10 point scale) most days of an average week

Exclusion Criteria:

* pregnant
* diagnosed by doctor with sleep apnea, facial or airways defect
* any facial or airways surgery that has changed snoring pattern.
* upper airways infection that requires antibiotics, cough suppressants, etc. in the last month
* use any continuous positive airway pressure (CPAP) device or dental appliance
* bed partner hearing impairment or defects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Snoring | 4 weeks

SECONDARY OUTCOMES:
Sleep Quality | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Littenberg, MD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States